CLINICAL TRIAL: NCT05836922
Title: Association Between Renal Regional Oxygen Saturation Measured by Near-InfraRed Spectroscopy and Postoperative Renal Failure After Lung Transplantation Surgery: A Pilot Study
Acronym: SO-AKI-TP
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM23_0007
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Lung Transplant; Complications; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Complications after lung transplantation are almost ubiquitous, among which postoperative acute renal failure may represent more than 50% of lung transplant patients and require extrarenal purification in 5 to 13% of cases.

Multiple factors are associated with postoperative acute renal failure. These factors can be classified into preoperative, intraoperative, and postoperative factors. While some postoperative complications are explained by donor and recipient factors, the literature suggests that certain intraoperative events represent modifiable or avoidable risk factors that could be targeted by therapeutic interventions to reduce the risk of postoperative acute renal failure. Some of these factors (intraoperative hemodynamic instability, significant bleeding or hypoxemia) can generate renal hypoxic aggression, alone or in combination. However, to date, there is no validated tool available at the patient's bedside during surgery to detect renal hypoxia or guide interventions to restore renal perfusion during surgery. Yet, as recent recommendations suggest, intraoperative renal protection is an important axis for improving the outcome of lung transplant patients, to the extent that the recommendations of Marczin et al. recommend the establishment of a renal prevention protocol for each patient. Without a tool to guide this plan intraoperatively, anesthesia teams can't establish a renal prevention protocol. This research aims to establish whether renal NIRS is a reliable tool for monitoring intraoperative renal hypoxic aggression predictive of postoperative renal failure.

Near-infrared spectroscopy (NIRS) is an optical technology that allows non-invasive measurement of tissue oxygen saturation. This technique is commonly used for intraoperative monitoring of cerebral perfusion in adults and children. Some studies have shown that regional renal oxygen saturation (renal rSO2) measured by NIRS during aortic-coronary bypass surgery under extracorporeal circulation (ECC) is correlated with renal venous oxygen saturation measured by catheterization. It is also associated with the risk of postoperative acute renal failure in patients undergoing cardiac surgery under ECC. However, there are no equivalent data in lung transplant patients, who frequently present with postoperative acute renal failure. In the available literature, no clear threshold of renal desaturation has been established. Because it is assumed that the depth of renal desaturation can be particularly deleterious, in addition to desaturation time, the investigator have chosen to retain in this project the integral of time and magnitude spent under a renal desaturation threshold, aggregated into a renal hypoxia index, during the intraoperative period.

The primary objective of this research is to demonstrate the usefulness of measuring the intraoperative renal hypoxia index in predicting the risk of early postoperative acute renal failure

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing a lung transplant (mono or bi-transplantation)
* Age >= 18 years
* Affiliated to the French social security system

Exclusion Criteria:

* Renal anatomical abnormality likely to induce a misleading NIRS signal: single kidney, polycystic kidney disease.
* Expression of opposition to participation in the research protocol.
* Hyperbilurbinemia > 17mmol/l
* Preoperative Extra Corporeal Membran Oxygenation (ECMO).
* Preoperative mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a lung transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Relation between renal hypoxia index and AKI | 5 days postoperative
  Early postoperative acute kidney injury (AKI) is determined by a KDIGO stage ≥ 1 occurring between the end of the surgery and the 5th postoperative day (the KDIGO stage is defined by the variation of serum creatinine and urine output according to The Kidney Disease Improving Global Outcomes (KDIGO) Working Group).
  The renal hypoxia index is expressed in %·min. It will be tested for several critical saturation thresholds: 70%, 65%, 60%, 55%, 50%. The threshold of 65% is selected for the main analysis based on the work of Ortega-Loubon, and the other thresholds will be tested in a secondary analysis.
  For the main analysis, the interest of the index will be demonstrated by comparing the means of this index between the group that developed AKI and the group that did not. In the secondary analysis, the interest of the index will be demonstrated by studying the performance of the index for the occurrence of AKI, by estimating the ROC curve and the area under the ROC curve.

SECONDARY OUTCOMES:
Relation between renal hypoxia index and renal replacment therapy | 5 days postoperative
  The use of renal replacement therapy during the 5 first postoperative days
Relation between renal hypoxia index and primary graft dysfuncion | 5 days postoperative
  Primary graft dysfunction based on ISHLT 2016 stadification
Relation between hypotension index and acute kidney injury | 5 days postoperative
  The hypotension index represent the time spent below 65mmHg of Mean Arterial Pressure (PAM) during the surgery is expressed in mmHg.min.Early postoperative acute kidney injury is determined by a KDIGO stage ≥ 1 occurring between the end of the surgery and the 5th postoperative day (the KDIGO stage is defined by the variation of serum creatinine and urine output according to The Kidney Disease Improving Global Outcomes (KDIGO) Working Group).

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — Assistance Publique Hopitaux De Marseille

IPD SHARING:
Plan to Share IPD: Undecided